CLINICAL TRIAL: NCT01746355
Title: Assessment and Treatment Patients With Atypical Facial Pain Trough Repetitive Transcranial Magnetic Stimulation
Acronym: EMTr-AFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Galhardoni, PhD student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: RG-01
Record Dates: First submitted 2012-11-27; First posted 2012-12-10 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Atypical Facial Pain or Atypical Odontalgia
Keywords: atypical facial pain; atypical odontalgia; repetitive transcranial magnetic stimulation; neuropathic pain; chronic pain; assessment
MeSH Terms: conditions — Neuralgia; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS-active (Active Comparator): patients undergoing of rTMS real
  Interventions: Procedure: rTMS
- rTMS-Sham (Sham Comparator): patients undergoing to placebo rTMS
  Interventions: Procedure: rTMS

INTERVENTIONS:
Procedure: rTMS — Patients undergoing of repetitive transcranial magnetic stimulation for treatment of AFP.

SUMMARY:
Atypical Facial Pain is a chronic condition and presents controversies during diagnostic and treatment, between specialist not have consensus about the pathophysiology. It is possible consider this entitie a potential neuropathic cause without pathological signs. It knows the repetitive transcranial magnetic presents good results in the treatment of chronic pain coditions. The aim this study is evaluated the thresholds and excitability cortical in patients with AFP and verify the patterns of improvement in pain for patients undergoing rTMS compared to controls, as well as the therapeutic response to neuromodulation procedures. This enroll 20 patients with DAF and 20 controls treated with rTMS (5 sessions) and evaluated through questionnaires (EDOF clinical record, McGill Pain Questionnaire, Visual Analogue Scale, Inventory of symptoms of neuropathic pain, neuropathic pain DN4 questionnaire, SF -36, brief pain inventory). At the end of the data will be statistically analyzed and expressed as mean and standard deviation, and analyzed by Student's t test, analysis of variance (ANOVA), Tukey-Kramer and Pearson correlation. The level of significance is 5%. The results will be published in journals indexed in the area both nationally and internationally and presented at conferences and scientific meetings.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill criteria of Atypical Facial Pain by International Headache Society
* Signed Term of Informed Consent

Exclusion Criteria:

* Trauma of Skull, epilepsy don't treated,
* Use of medications decrease the seizure threshold
* Patients in use of drugs, how cocaine and alcohol
* neurosurgical clips, pacemakers, increased intracranial pressure (risk of sequelae after seizure)
* Pregnant or lacting women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Baselin of Pain | base line (moment of inclusion) and end of each session rTMS (4X in three months)
  Assessing by verbal analog scale (VAS)

SECONDARY OUTCOMES:
Excitability cortical | baseline (in the moment of inclusion) and end of each session of rTMS (4X in three months)
  Changes in the measure of excitability cortical

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HC/FMUSP), São Paulo, São Paulo, Brazil